CLINICAL TRIAL: NCT06093308
Title: A Phase 1, Open-label, Single-and Multiple-dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of JT001 Administered Orally in Elderly Chinese Subjects With Underlying Diseases
Brief Title: A Study in Elderly Chinese Subjects With Underlying Diseases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Vinnerna Biosciences Co., Ltd. (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: JT001-017-I
Record Dates: First submitted 2023-09-25; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Elderly Subjects With Underlying Diseases
MeSH Terms: interventions — GS-621763

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Elderly subjects (Experimental): elderly subjects with underlying diseases.
  Interventions: Drug: Deuremidevir Hydrobromide Tablets

INTERVENTIONS:
Drug: Deuremidevir Hydrobromide Tablets — Multiple administration, oral administration after meals, D1: 0.6g, twice a day; D2-D5: 0.3g, twice a day; D6: 0.3g, administered once in the morning
  Other Names: JT001

SUMMARY:
Evaluate the safety and tolerability of oral JT001 tablets in elderly subjects with underlying diseases.

Evaluate the pharmacokinetic characteristics of JT001 tablets orally administered to elderly subjects with underlying diseases.

Explore the drug drug interactions between JT001 tablets and some drugs in elderly subjects with underlying diseases who have been orally administered multiple times.

DETAILED DESCRIPTION:
The open-label, single-center phase I study to evaluate the safety, tolerability, and pharmacokinetics of JT001 single-and multiple-dose administered orally in elderly subjects with underlying diseases.Approximately 16 to 18 elderly subjects will be enrolled aging beyound 60 years.

All subjects received JT001, oral administration after meals, D1: 0.6g, twice a day; D2-D5: 0.3g, twice a day; D6: 0.3g, administered once in the morning.Blood samples will be collected at times sufficient to adequately define the pharmacokinetics of JT001 active metabolite(116N-1) in elderly groups.The steady-state trough concentration of therapeutic drug monitoring (TDM) for the basic medication of the subjects will be collected as well.

Subjects will be admitted to the phase I clinical trial ward 2 days before administration (D-2) and will not be allowed to leave until all examinations and assessments are completed on day 8. Telephone follow-up will be performed on day 12 (±1 day).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 60 years old, regardless of gender;
2. Weight: Male ≥ 50 kg, female ≥ 45 kg; Body mass index (BMI) within the range of 18-30 kg/m2 (including 18 and 30);
3. Subjects suffer from chronic basic diseases and have stable disease control (such as well controlled hypertension, hyperlipidemia, diabetes, etc.);
4. At least 2 weeks before enrollment, the treatment plan for chronic underlying diseases of the subjects has not been adjusted, and the usage, dosage, and duration of the treatment drugs remain unchanged;
5. During the study period, the subjects were willing to discontinue non essential concomitant medications or health products (excluding essential treatment drugs for chronic underlying diseases of the subjects, and the specific drugs and health products were determined by the researchers and specialist doctors in consultation);
6. The results of vital signs, physical examinations, routine laboratory tests (blood routine, blood biochemistry, urine routine, coagulation function, etc.), 12-lead electrocardiogram, chest X-ray, abdominal ultrasound, etc. are normal or abnormal, but the researchers determine that they are related to age and chronic diseases. After enrollment, the safety risk of the subjects is low and does not affect the study observation indicators;
7. Those who understand the research procedures and methods, voluntarily participate in this study, and sign an informed consent form in writing.

Exclusion Criteria:

1. Individuals with a known history of allergies, allergic diseases, or allergic constitutions to the research formulation, any of its components, or related preparations;
2. Any surgical situation or condition that may significantly affect the absorption, distribution, metabolism, and excretion of drugs, or any surgical situation or condition that may pose a hazard to the participants in the study, such as a history of gastrointestinal surgery (gastrectomy, gastrointestinal anastomosis, intestinal resection, etc.), a history of gastroenteritis, gastrointestinal ulcers, gastrointestinal bleeding, history of malignant tumors, etc. (excluding cholecystectomy);
3. Those who have experienced the following conditions within 3 months prior to the administration of the study drug: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass grafting, congestive heart failure, severe arrhythmia, cerebrovascular accidents, including transient ischemic attacks;
4. Individuals who have experienced blood loss of ≥ 400 mL within the first 3 months of enrollment;
5. Individuals who have participated in clinical research on other drugs or medical devices within the first 3 months of being selected;
6. Drink alcohol at least twice a day or more than 14 times a week within 6 months before selection, or indulge in excessive drinking (one drink is defined as 125 mL of wine, 220 mL of beer or 50 mL of Baijiu; excessive drinking is defined as five or more drinks within about 2 hours);
7. Individuals with a history of drug use or positive drug abuse screening;
8. Those who smoke more than 10 cigarettes per day within the first 6 months of enrollment;
9. Positive individuals for hepatitis B surface antigen (HBsAg), HCV antibody, Treponema pallidum antibody, and HIV antibody;
10. Researchers believe that there are other factors that are not suitable for participating in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-07-12 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
The severity of SAE | From Day 1(first dose) to Day12
  The severity of SAE
The Number of participants with SAE | From Day 1(first dose) to Day12
  The Number of participants with SAE
The severity ofclinical symptoms abnormalities(e.g.,Dizziness, headache, nausea, abdominal pain, fatigue, drowsiness） | From Day 1(first dose) to Day12
  The severity ofclinical symptoms abnormalities(e.g.,Dizziness, headache, nausea, abdominal pain, fatigue, drowsiness）
The Number of participantswith abnormal clinical symptoms(e.g.,Dizziness, headache, nausea, abdominal pain, fatigue, drowsiness） | From Day 1(first dose) to Day12
  The Number of participantswith abnormal clinical symptoms(e.g.,Dizziness, headache, nausea, abdominal pain, fatigue, drowsiness）
The severity of vital signs abnormalities | From Day 1(first dose) to Day12
  The severity of Pulse abnormalities
The Number of participantswith abnormal vital signs | From Day 1(first dose) to Day12
  The Number of participantswith abnormal Pulse
The severity of vital signs abnormalities | From Day 1(first dose) to Day12
  The severity of blood pressure abnormalities
The Number of participantswith abnormal vital signs | From Day 1(first dose) to Day12
  The Number of participantswith abnormal blood pressure
The severity of vital signs abnormalities | From Day 1(first dose) to Day12
  The severity of respiration abnormalities
The Number of participantswith abnormal vital signs | From Day 1(first dose) to Day12
  The Number of participantswith abnormal respiration
The severity of vital signs abnormalities | From Day 1(first dose) to Day12
  The severity of body temperature abnormalities
The Number of participantswith abnormal vital signs | From Day 1(first dose) to Day12
  The Number of participantswith abnormal body temperature
The severity of vital signs abnormalities | From Day 1(first dose) to Day12
  The severity of abnormal physical examinations findings
The Number of participantswith abnormal physical examinations findings | From Day 1(first dose) to Day12
  The Number of participantswith abnormal physical examinations findings
The severity of abnormal laboratory tests results | From Day 1(first dose) to Day12
  The severity of abnormal laboratory tests results
The Number of participantswith abnormal laboratory tests results | From Day 1(first dose) to Day12
  The Number of participantswith abnormal laboratory tests results
The severity of electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The severity of Heart rate abnormalities
The Number of participants with electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The Number of participants with Heart rate abnormalities
The severity of electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The severity of PR interval abnormalities
The Number of participants with electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The Number of participants with PR interval abnormalities
The severity of electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The severity of QRS interval abnormalities
The Number of participants with electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The Number of participants with QRS interval abnormalities
The severity of electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The severity of QT interval abnormalities
The Number of participants with electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The Number of participants with QT interval abnormalities
The severity of electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The severity of QTcF abnormalities
The Number of participants with electrocardiogram (ECG) abnormalities | From Day 1(first dose) to Day7
  The Number of participants with QTcF abnormalities

SECONDARY OUTCOMES:
The Cmax of the main metabolite 116-N1 of JT001; | Day 1/Day 5 and Day 6 after first dose
  area under curve from time zero to infinity
The AUC0-t of the main metabolite 116-N1 of JT001; | Day 1/Day 5 and Day 6 after first dose
  area under curve from time zero to infinity
The AUC0-inf of the main metabolite 116-N1 of JT001; | Day 1/Day 5 and Day 6 after first dose
  area under curve from time zero to infinity

OTHER OUTCOMES:
The steady-state trough concentration of therapeutic drug monitoring (TDM) for the basic medication of the subjects. | Day 2 and Day 1before first dose and Day 6/Day 7/Day 8 after first dose
  The steady-state trough concentration of therapeutic drug monitoring (TDM)

CONTACTS AND LOCATIONS:
Overall Officials: Huiyu Lan, Project Director, Study Director — Shanghai Vinnerna Biosciences Co., Ltd.
Locations (1):
- Shanghai Xuhui Central Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Undecided